CLINICAL TRIAL: NCT06654934
Title: Prednisolone for 12 Versus 6 Months to Treat Pulmonary Sarcoidosis: a Randomized Trial
Brief Title: Prednisolone for 12 Versus 6 Months to Treat Pulmonary Sarcoidosis
Acronym: DURASARC
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sahajal Dhooria, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pulm-962
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Sarcoidosis
Keywords: granulomatous disease; interstitial lung disease; diffuse lung disease; tuberculosis; steroid; ILD
MeSH Terms: conditions — Sarcoidosis; Lung Diseases, Interstitial; Tuberculosis | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short duration (Active Comparator): 6-month prednisolone (shorter treatment)
  Interventions: Drug: Prednisolone
- Long duration (Active Comparator): 12-month prednisolone (longer treatment)
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — An initial dose of 40 mg/day will be administered for 1 week, followed by 30 mg/day for 1 week, 20 mg/day for 6 weeks, 15 mg/day for 4 weeks, 10 mg/day for 8 weeks, 5 mg/day for 4 weeks, 2.5 mg/day for 2 weeks after which the drug will be discontinued (cumulative prednisolone dose, 2485 mg).
  Arms: Short duration
Drug: Prednisolone — An initial dose of 40 mg/day will be administered for 1 week, followed by 30 mg/day for 1 week, 20 mg/day for 6 weeks, 15 mg/day for 4 weeks, 10 mg/day for 14 weeks, 5 mg/day for 24 weeks, 2.5 mg/day for 2 weeks after which the drug will be discontinued (cumulative prednisolone dose, 3605 mg).
  Arms: Long duration

SUMMARY:
In this study, the efficacy and safety of treating pulmonary sarcoidosis with 12 months vs. 6 months of prednisolone will be compared. The hypothesis is that longer treatment DURAtion would be more effective in preventing treatment failure or early relapse in SARCoidosis (DURASARC trial). The premise of this hypothesis is that even small doses of prednisolone given over longer periods can effectively suppress disease activity in sarcoidosis without a significant increase in adverse effects.

DETAILED DESCRIPTION:
Sarcoidosis is an idiopathic disorder that manifests with granulomatous inflammation affecting several organs, but most commonly the lungs and mediastinal lymph nodes. When asymptomatic or minimally symptomatic, it does not require regular pharmacologic treatment. Organ dysfunction or impaired quality of life trigger the introduction of immunosuppressive therapy. Glucocorticoids are the first-line drugs for this purpose. Different glucocorticoids have been studied in the past, but prednisone/prednisolone is the most used agent. Evidence is sparse on the ideal glucocorticoid regimen to treat patients with sarcoidosis. A recent randomized controlled trial (RCT) named the SARCORT study found that a 6-month prednisolone regimen using an initial dose of 40 mg/day was not superior to one that initiated with a daily dose of 20 mg. The appropriate duration of glucocorticoid treatment for treating newly diagnosed patients with sarcoidosis is unknown.

The treatment duration of 6 months in the SARCORT study was at the shorter end of the suggested range (6-24 months). There was a high (45%) overall relapse incidence which was proposed to be due to the shorter duration of treatment. In contrast, a study with a glucocorticoid treatment duration of one year described a 13% relapse rate. In another study, significantly better results were observed in patients who had received prolonged treatment for 4 years or more.

In this study, the aim is to compare the efficacy and safety of treating pulmonary sarcoidosis with 12 months vs. 6 months of prednisolone. The hypothesis is that longer treatment DURAtion would be more effective in preventing treatment failure or early relapse in SARCoidosis (DURASARC trial). The premise of this hypothesis is that even small doses of prednisolone given over longer periods can effectively suppress disease activity in sarcoidosis without a significant increase in adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Computed tomography of the chest consistent with a diagnosis of sarcoidosis of the lung/mediastinal lymph nodes
* Diagnosis of sarcoidosis made on cytological or histological samples
* Having significant symptoms requiring immunosuppressive treatment and/or having reduced lung function (defined as forced vital capacity or forced expiratory volume in one second (FEV1) less than 80% predicted) or an extrapulmonary manifestation of the disease requiring treatment with low-medium dose glucocorticoids
* Onset of symptoms within two years of study entry

Exclusion Criteria:

* Pregnant or lactating women
* Subjects having any manifestation requiring high dose steroid treatment (this includes symptomatic neurosarcoidosis, life threatening cardiac sarcoidosis, vision threatening posterior uveitis or other forms of vision threatening ocular sarcoidosis)
* Having absolute contraindication for prednisone (this includes untreated glaucoma, uncontrolled diabetes mellitus, untreated infections, untreated severe psychiatric disorders)
* Unwilling to participate in the study
* Having received glucocorticoids (prednisolone equivalent >15 mg/day) for more than three weeks in the preceding year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Relapse or treatment failure | 12 months
  Proportion of subjects with a relapse (worsening after 4 weeks of stopping treatment) or treatment failure (worsening during treatment or within 4 weeks of stopping treatment requiring an increase in the treatment intensity) in the study groups. Worsening is defined as persistent (≥2 weeks) worsening of cough and/or dyspnea, and one or more of the following: a) worsening of lung function (≥5-point reduction in percentage-predicted FVC or FEV1), or b) increase in the chest radiograph abnormalities due to sarcoidosis.

SECONDARY OUTCOMES:
Treatment response | 12 months
  Proportion of subjects with good or fair treatment response between the study groups defined as:
  Good response: Resolution (no symptoms attributable to sarcoidosis, a normal chest radiograph, and normal lung function with normal laboratory parameters related to the initial treatment-requiring indication) or improvement (improvement in respiratory symptoms with either (a) decrease in radiological abnormalities, or (b) a ≥5-point increase in the percentage-predicted FVC or FEV1 from the baseline, or (c) both, with no worsening on imaging or spirometry along with normal/stable laboratory parameters related to the initial treatment-requiring indication) with treatment.
  Fair response: Stabilization (any reduction in symptoms along with stable radiological abnormalities, and less than a 5-point change in the percentage-predicted FVC and FEV1 along with normal/stable lab parameters) of disease during treatment.
Sarcoidosis health related quality of life | 12 months
  Sarcoidosis health related quality of life will be assessed using the King's Sarcoidosis Questionnaire (KSQ). KSQ is a validated multidomain instrument used to assess QoL of patients with sarcoidosis. The domains include: general health (GH), lung, medication, skin and eyes. The questionnaire consists of 29 items (general health: 10, lung: 6, medication: 3, skin: 3, eyes: 7) that assess the disability that the symptoms in various domains have posed on the patient's day-to-day activities in the past week. Each item is rated on a 7-point Likert scale from 1 (all of the time) to 7 (none of the time). The KSQ module and overall (total) scores are finally transformed to a range of 0-100 [(actual score - lowest possible score/range) ×100], where higher scores represent better health status. A minimal clinically important difference (MCID) of 8 for the KSQ GH and of 4 for the KSQ lung have been proposed in a study of 271 subjects.
Forced vital capacity | 12 months
  Mean change in forced vital capacity assessed using spirometry between the study groups. Spirometry will be performed according to the ATS/ERS guidelines using an ultrasonic flow sensor spirometer (NDD Medizintechnik AG, Zurich, Switzerland) and will be expressed in liters.
Adverse effects | 12 months
  Proportion of subjects having glucocorticoid-related adverse effects will be recorded including weight gain, Cushingoid features, infections, skin thinning, ecchymosis, cataracts, increased intraocular pressure, hypertension, gastritis, osteoporosis, myopathy, mood disorder, psychosis, memory impairment, hyperglycemia, and others.
Time to relapse or treatment failure | 12 months
  Mean time to relapse (worsening after 4 weeks of stopping treatment) or treatment failure (worsening during treatment or within 4 weeks of stopping treatment requiring an increase in the treatment intensity) in the study groups. Worsening is defined as persistent (≥2 weeks) worsening of cough and/or dyspnea, and one or more of the following: a) worsening of lung function (≥5-point reduction in percentage-predicted FVC or FEV1), or b) increase in the chest radiograph abnormalities due to sarcoidosis
Sarcoidosis-associated fatigue | 12 months
  Sarcoidosis-associated fatigue will be assessed using the Fatigue assessment scale (FAS). FAS is a questionnaire with ten items, with five ques¬tions for physical fatigue and five questions reflecting mental fatigue.25 The questionnaire is self-completed by patients and all question¬naire items are rated on a five-point Likert scale (1, never to 5, always). The response scores are sum¬mated to get a total score, which ranges from 10- 50. FAS scores ≥22 and ≥35 imply fatigue and severe fatigue respectively.26 A four-point change in FAS scores after treatment is considered clinically significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study, including deidentified participant data and related documents, including the protocol, statistical analysis plan, and informed consent form, will be made available to qualified researchers after the publication of the manuscript upon reasonable request made to the Principal Investigator (S. Dhooria) after the publication of the primary manuscript.
Supporting Information: Study Protocol, SAP
Time Frame: Anticipated: 31-Dec-2026 till indefinite